CLINICAL TRIAL: NCT06696326
Title: A Multicenter Study Evaluating the Diagnostic Value of 68Ga-MY6349 PET/CT for Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XMYY-2024KY171
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Positron-Emission Tomography(PET); Prostate Cancer; Trophoblast Cell Surface Antigen 2
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-MY6349 (Experimental): Each subject receives a single intravenous injection of 68Ga-MY6349 and undergoes PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: standard-of-care imaging 68Ga-MY6349 and 68Ga-PSMA-11

INTERVENTIONS:
Diagnostic Test: standard-of-care imaging 68Ga-MY6349 and 68Ga-PSMA-11 — Each subject receives a single intravenous injection of standard-of-care imaging radiopharmaceuticals 68Ga-MY6349 and 68Ga-PSMA-11, and undergoes PET/CT imaging within the specified time.

SUMMARY:
The main objective of this research is to develop and evaluate new PET imaging agents with high sensitivity and specificity for prostate cancer and other aggressive tumors. Specifically, the research focuses on improving upon existing prostate cancer imaging methods, such as PSA tests and PSMA PET/CT, which have limitations in sensitivity, specificity, and the ability to provide comprehensive tumor information，and aims to create a novel PET probe targeting Trop2, an antigen highly expressed in multiple cancer types, to enable in vivo, whole-tumor assessment. This would support early diagnosis, more precise staging, and effective monitoring of cancer therapy.

DETAILED DESCRIPTION:
Prostate cancer is the second most common cancer in men and the fifth leading cause of male cancer-related death. Incidence rates are higher in developed countries (37.5 per 100,000) compared to developing countries (11.3 per 100,000), with similar patterns in mortality rates. Currently, approximately 10 million men are diagnosed with prostate cancer worldwide, with over 400,000 deaths annually. By 2040, annual mortality is projected to reach over 800,000. Detection methods for prostate cancer include digital rectal examination, serum prostate-specific antigen (PSA), ultrasound, CT, MRI, and bone scans. While helpful, these methods have limitations, particularly in early detection, biochemical recurrence, and post-treatment assessment. Hence, there is a pressing need for sensitive and specific diagnostic agents capable of detecting and localizing tumors and small metastases for accurate diagnosis, staging, and recurrence assessment. In recent years, PET molecular imaging, which visualizes biochemical metabolism and specific target expression, has provided valuable insights into tumor biology. Prostate-specific membrane antigen (PSMA), a type II glutamate carboxypeptidase produced by prostate epithelial cells, is highly expressed in prostate cancer and its metastases, with minimal expression in other normal tissues (e.g., intestines, brain, kidneys) at levels significantly lower than in cancer tissues. This specificity makes PSMA a crucial target for prostate cancer imaging. Two PET radiotracers, 68Ga-PSMA-11 and 18F-DCFPyL, are now FDA-approved in the United States for imaging prostate cancer, particularly for detecting recurrence. While these tracers offer high sensitivity and specificity, there are still some limitations. On the one hand, despite the high sensitivity of PSMA PET/CT, false positives can occur due to benign prostate hyperplasia, prostatitis, or other non-cancerous conditions that may also express PSMA. Additionally, some low-grade or small tumors, as well as neuroendocrine-differentiated prostate cancers, may not express sufficient PSMA, resulting in false negatives. On the other hand, PSMA PET/CT primarily detects PSMA-expressing tissues but does not provide information on other tumor biological characteristics, which may limit its utility in therapeutic decision-making and prognostic assessment. Trophoblast cell surface antigen 2 (Trop2) is another promising target, highly expressed in various cancers. Antibody-drug conjugates (ADCs) targeting Trop2 have demonstrated clinical success in treating advanced triple-negative breast cancer, HR+/HER2- breast cancer, and urothelial carcinoma, offering new options for patients with late-stage cancers resistant to multiple treatments. Since ADC efficacy is closely linked to antigen expression, Trop2 levels serve as a critical marker for predicting Trop2-ADC effectiveness. Currently, Trop2 detection is limited to immunohistochemical staining of biopsy samples, which reflects only local expression and cannot represent Trop2 levels across entire tumors or metastases. Thus, a comprehensive, in vivo, dynamic method for Trop2 expression detection is needed. Our research team has successfully developed a Trop2-specific nanobody and constructed a novel Trop2 PET probe labeled with 68Ga. This probe effectively identifies Trop2 expression in different tumor models, showing favorable pharmacokinetics and tumor uptake. Initial clinical research suggests that 68Ga-MY6439 demonstrates higher uptake in prostate cancer than 18F-FDG and 68Ga-PSMA-11 PET/CT, detecting more lesions in certain cases with increased diagnostic sensitivity. Therefore, beyond patient selection for Trop2-ADC therapy, Trop2-targeted PET probes have potential as broad-spectrum imaging agents for malignancies, aiding in the diagnosis, staging, and therapeutic monitoring of aggressive cancers, potentially overcoming limitations seen with 18F-FDG and 68Ga-PSMA-11 PET/CT in certain tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with initial diagnosis of prostate cancer, or patients with biochemical recurrence after radical prostatectomy or radical radiotherapy.
2. Estimated survival time >3 months, as determined by a physician.
3. Willing to sign the informed consent form voluntarily and able to comply with the study protocol.

Exclusion Criteria:

1. Individuals unable to tolerate intravenous administration (e.g., history of needle or blood phobia).
2. Patients deemed unsuitable by researchers or unable to complete PET or other imaging examinations due to specific conditions, such as claustrophobia or radiophobia.
3. Individuals with occupational exposure to radiation.
4. Patients with severe diseases affecting the heart, kidneys, lungs, vascular, neurological, or mental systems, immune deficiency disorders, or hepatitis/cirrhosis.
5. Other conditions that researchers deem unsuitable for participation in the study.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 2 years
  The sensitivity, specificity, and accuracy of 68Ga-MY6349 and 68Ga-PSMA-1PET/CT were calculated and compared to evaluate the diagnostic accuracy.

SECONDARY OUTCOMES:
Number of lesions | 2 years
  The numbers of positive primary and metastatic lesions of 68-MY6349 PET/CT and 68Ga-PSMA-11 PET/CT were recorded by visual interpretation.
SUV | 2 years
  Standardized uptake value (SUV) of 68-MY6349 PET/CT and 68Ga-PSMA-11 PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No